CLINICAL TRIAL: NCT04501601
Title: The Effect of Consuming on Body Composition and Blood Biochemistry Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-039-A
Record Dates: First submitted 2020-08-02; First posted 2020-08-06 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Gut Microbiota
Keywords: Anthropometric index; Biochemical items
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: weight loss program kit (Experimental): weight loss program kit
  Interventions: Dietary Supplement: Fruit and vegetable solid drink

INTERVENTIONS:
Dietary Supplement: Fruit and vegetable solid drink — weight loss program supplement

SUMMARY:
To assess the effect of consuming on body composition and blood biochemistry index

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 20 and 60 years old
* Body mass index (BMI) ≥ 24 (kg/m^2) or body fat mass: male > 25%, female > 30%
* Prohibitions on other nutritional supplements (probiotics and prebiotics) before two weeks of the study
* Abidance by the similar diet and exercise habits over the study.

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Menopausal woman
* Diabetes mellitus
* Implementation in weight loss programs before a half year of this study
* Metabolic disorders
* Kidney diseases
* Liver diseases
* Cardiovascular diseases
* Nervous system diseases
* Gastrointestinal diseases
* Heavy drinking or constant drug use.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The change of body fat mass | Change from Baseline body fat mass at 2 months
  The body fat mass (kg) was assessed by InBody770.
The change of Triglyceride | Change from Baseline triglyceride at 2 months
  Venous blood was sampled to measure concentrations of Triglyceride
The change of Total cholesterol | Change from Baseline total cholesterol at 2 months
  Venous blood was sampled to measure concentrations of Total cholestrol
The change of HDL-cholesterol | Change from Baseline HDL-cholesterol at 2 months
  Venous blood was sampled to measure concentrations of HDL-cholestrol
The change of LDL-cholesterol | Change from Baseline LDL-cholesterol at 2 months
  Venous blood was sampled to measure concentrations of LDL-cholestrol
Fecal microbiome analysis | Change from Baseline Fecal microbiome at 2 months
  Firmicutes, Bacteroidetes, Lactobucillius, and A. muciniphila were quantified by quantitative PCR.
The change of body mass index (BMI) | Change from Baseline body mass index at 2 months
  BMI is a measurement of a person's leanness or corpulence based on their height and weight, and is intended to quantify tissue mass.The body mass index (BMI, kg/m^2) and body mass (kg) were assessed by InBody770.
The change of body fat percentage | Change from Baseline body fat percentage at 2 months
  The body fat percentage (%) was assessed by InBody770
The change of visceral fat | Change from Baseline visceral fat at 2 months
  The visceral fat (10 cm^2) was assessed by InBody770.

SECONDARY OUTCOMES:
The change of fasting glycemia | Change from Baseline fasting glycemia at 2 months
  Venous blood was sampled to measure concentrations of fasting glycemia
The change of aspartate aminotransferase | Change from Baseline aspartate aminotransferase at 2 months
  Venous blood was sampled to measure concentrations of aspartate aminotransferase
The change of alanine aminotransferase | Change from Baseline alanine aminotransferase at 2 months
  Venous blood was sampled to measure concentrations of alanine aminotransferase
The change of albumin | Change from Baseline albumin at 2 months
  Venous blood was sampled to measure concentrations of albumin
The change of creatinine | Change from Baseline creatinine at 2 months
  Venous blood was sampled to measure concentrations of creatine
The change of uric acid | Change from Baseline uric acid at 2 months
  Venous blood was sampled to measure concentrations of uric acid
The change of white blood cell | Change from Baseline white blood cell at 2 months
  Venous blood was sampled to measure concentrations of white blood cell

CONTACTS AND LOCATIONS:
Overall Officials: Bo-Han Wu, Principal Investigator — Study Principal Investigator
Locations (1):
- National Pingtung University of Science and Technology, Pingtung City, Neipu Township, Taiwan